CLINICAL TRIAL: NCT06765447
Title: EFFECT of USE of DIODE LASER and 3% NaOCl for HEMOSTASIS in DIRECT PULP CAPPING on OUTCOME in MILD and MODERATE PULPITS:A PROSPECTIVE CLINICAL STUDY.
Brief Title: EFFECT of USE of DIODE LASER and 3% NaOCl for HEMOSTASIS in DIRECT PULP CAPPING on OUTCOME in MILD and MODERATE PULPITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr. Varsha
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2023-06

CONDITIONS: HEMOSTASIS; DIRECT PULP CAPPING
MeSH Terms: interventions — Hemostasis; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3% NaOCl (Active Comparator): after pulp exposure bleeding was control by placing a cotton pellet soaked with 3%NaOCl over the pulpal wound upto 1 minutes.If hemostasis was not achieve with in 1mins we again use soaked cotton pellet of 3% NaOCL for another 1 mint until the hemostasis acheived. Tooth with excessive uncontrollable bleeding even after 5 mins was excluded from the study
  Interventions: Procedure: hemostasis with 3% NaOCl in direct pulp capping; Procedure: hemostasis with diode laser in direct pulp capping
- diode laser (Experimental): Hemostasis was achieved by exposure to Primo dental diode laser by medency (980 nm), at 0.5 W(medency Primo laser) .During laser application patients, operator and assistant were asked to wear protective eye shields.The laser energy of wavelength 980 nm introduced to the exposure site through a 400 µm optical fiber in a non contact mode for 2-3 seconds at exposure site for three times at 10s time interval to achieve complete hemostasis.For disinfection same diode laser of wavelength 980nm with energy set at 1W used in non contact mode in circular motion in the cavity
  Interventions: Procedure: hemostasis with 3% NaOCl in direct pulp capping; Procedure: hemostasis with diode laser in direct pulp capping

INTERVENTIONS:
Procedure: hemostasis with 3% NaOCl in direct pulp capping — after pulp exposure bleeding was control by placing a cotton pellet soaked with 3%NaOCl over the pulpal wound upto 1 minutes.If hemostasis was not achieve with in 1mins we again use soaked cotton pellet of 3% NaOCL for another 1 mint until the hemostasis acheived. Tooth with excessive uncontrollable bleeding even after 5 mins was excluded from the study; however, definite treatment was provided to the patient.The time used to control bleeding was recorded for each tooth by using stop watch.Once hemostasis is achieved, exposed pulp was capped with biodentine.
Procedure: hemostasis with diode laser in direct pulp capping — Hemostasis was achieved by exposure to Primo dental diode laser by medency (980 nm), at 0.5 W(medency Primo laser) .During laser application patients, operator and assistant were asked to wear protective eye shields.The laser energy of wavelength 980 nm introduced to the exposure site through a 400 µm optical fiber in a non contact mode for 2-3 seconds at exposure site for three times at 10s time interval to achieve complete hemostasis.For disinfection same diode laser of wavelength 980nm with energy set at 1W used in non contact mode in circular motion in the cavity .Biodentine was used as pulp capping agent.

SUMMARY:
Goal of this prospective clinical study is evaluate the effect of use of diode laser and 3% NaOCl for hemostasis in direct pulp capping on outcome in mild and moderate pulpitis Population includes systemically healthy patient of age 18-45 years with extremely deep carious lesion in mandibular molar with normal periapical structure exibiting symptoms of mild and moderate pulpits .Clinical outcome assessed at 1 week and 3month by using electric pulp testing and cold test radiographic outcome will be assessed using periapical index scoring system at 6 and 12 months follow up period.

DETAILED DESCRIPTION:
Rationale: - Preservation of pulp vitality is a critical factor in long-term tooth survival. In deep carious lesion, vital pulp therapy procedures in the form of direct pulp capping is more conservative treatment strategy. When applied to dental tissues lasers have shown their potential to increase healing, control hemorrhage, stimulate dentinogenesis and preserve vitality of the dental pulp. Laser amplifies the healing process by stimulation of cell regeneration and is capable of inducing the odontoblasts for laying down tertiary dentine and forming a dentine bridge. Diode laser has great penetration, eliminate microorganism and has been shown to reduce post operative pain (Genc Sen, O.et al).Iraj Yazdanfar et al. evaluated the efficiency of diode 808-nm laser combined with Theracal LC in direct pulp capping performed on the caries-exposed pulps of permanent teeth and radiographically compared the thickness of dentin bridge formed for a 6-month follow-up. They found favorable results but recommended further studies with larger sample sizes, longer follow-up periods, and different capping material are needed to prove the effectiveness of the diode laser.

AIM & OBJECTIVES- To evaluate the effect of use of diode laser and 3% NaOCl for hemostasis in Direct Pulp Capping in mild and moderate pulpitis on success and survival.

Primary objective-To determine the success rate and survival of diode laser and sodium hypoclorite as hemostatic agent in direct pulp capping with biodentine, based on clinical findings at 1week,3 months and both clinical and radiographic findings at 6 and 12 months.Secondary objective-To assess the post operative pain from Day 1 to Day 7 post treatment(NRS score).

Participants:

Inclusion Criteria: -Healthy patients (ASA I ).Patients falling in the age group of 18-45 years.Unrestored Permanent mandibular posterior teeth.Extremely deep caries are defined as radiographic evidence of caries penetrating the entire thickness of the dentine with certain pulp exposure. In extremely deep lesions, the demineralized process extends the entire thickness of the dentine. (L.BJORNDAL et al.2019)Only occlusal pulp exposure due to caries.Vital teeth with signs and symptoms of mild and moderate pulpitis- Mild pulpitis Heightened and lengthened reaction to cold, warmth and sweet stimuli that can last up to 20 s but then subsides, possibly percussion sensitive. According to the histological situation that fits these findings, it would be implied that there is limited local inflammation confined to the crown pulp (W. J. Wolters et al.) Moderate pulpitis- Clear symptoms, strong, heightened and prolonged reaction to cold, which can last for minutes, possibly percussion sensitive and spontaneous dull pain that can be more or less suppressed with pain medication According to the histological situation that fits these findings, it would be implied that there is extensive local inflammation confined to the crown pulp (W. J. Wolters et al.).Exposure size 0.5 to 1 mm.

Exclusion Criteria: -No pulp exposure after caries excavation.No bleeding after pulp exposure.Participants who will not signed the written consent form.Patient with PAI score >2.Severe pulpits-There are any clinical symptoms of Severe spontaneous pain and clear pain reaction to warmth and cold stimuli, often, sharp to dull throbbing pain, patients have trouble sleeping because of the pain (gets worse when lying down). Tooth is very sensitive to touch and percussion.Evidence of internal or external resorption, calcified canals, as assessed by radiographic examination.Patients with periodontal disease, swelling and sinus tract.A positive history of antibiotic use within 1 month and analgesic use within week before the treatment.

Sample size: - 64 in one group Methods: - • The teeth were evaluated by periapical radiographs, periodontal probing, percussion test, and sensibility assessment with cold test and electric pulp test.All periapical radiographs were exposed by using constant kVP, mA, and exposure time (70 KVP, 8 mA, and 0.8 sec.).The tooth was anesthetized using lidocaine 2% with epinephrine 1:80,000 and subsequently isolated using rubber dam.The tooth was disinfected by scrubbing with 2% chlorhexidine and 75% isopropyl alcohol. Round diamond bur and high-speed handpiece with copious water irrigation was used to remove carious enamel and further round bur with low-speed handpiece was used to remove carious dentin.After pulp exposure, tooth was randomly allocated to one of the study groups for hemostasis achievement.To avoid selection bias,the randomization for diode laser and 3% NaOCl was done after pulp exposure .This was involve picking a closed envelope containing the instruction to either use NaOCl 3% or diode laser for hemostasis by an investigator who is not the part of study.

In GROUP 1,Hemostasis was achieved by exposure to Primo dental diode laser by medency (980 nm), at 0.5 W(medency Primo laser) .During laser application patients, operator and assistant were asked to wear protective eye shields.The laser energy of wavelength 980 nm introduced to the exposure site through a 400 µm optical fiber in a non contact mode for 2-3 seconds at exposure site for three times at 10s time interval to achieve complete hemostasis.For disinfection same diode laser of wavelength 980nm with energy set at 1W used in non contact mode in circular motion in the cavity .Biodentine was used as pulp capping agent.

In GROUP 2, after pulp exposure bleeding was control by placing a cotton pellet soaked with 3%NaOCl over the pulpal wound upto 1 minutes.If hemostasis was not achieve with in 1mins we again use soaked cotton pellet of 3% NaOCL for another 1 mint. Tooth with excessive uncontrollable bleeding even after 5 mins was excluded from the study; however, definite treatment was provided to the patient.The time used to control bleeding was recorded for each tooth by using stop watch.Once hemostasis is achieved, exposed pulp was capped with biodentine.Biodentine (Septodont, Saint-Maur-des-Fosses, France) aa was mixed according to manufacturer's instructions and applied directly onto the exposed pulpal site in 1- 2mm layer thickness. After 12-15 mins when Biodentine sets, application of RMGIC liner was done. This was followed by etching with 37% phosphoric acid for 15 seconds and rinsing with water. The cavity was then air dried and bonding agent was applied which was cured for 20 seconds. The cavity was then restored with composite using incremental technique FOLLOW UP:The patients were recalled periodically at 1 week, 3months, 6 months and 12 months after the direct pulp capping procedure for clinical evaluation (post operative sensitivity, pain, tenderness, vitality) and at 6 months and 12 months for radiographic (widening of periodontal ligament space and periapical radiolucency) evaluation.

ELIGIBILITY:
Inclusion Criteria:

1.Healthy patients (ASA I ).2.Patients in the age group of 18-45 years.Unrestored permanent mandibular posterior teeth.3.Extremely deep caries defined as radiographic evidence of caries penetrating the entire thickness of the dentine with certain pulp exposure. In extremely deep lesions, the demineralized process extends the entire thickness of the dentine, which perhaps excludes these cases from selective caries removal and a strategy based on avoiding pulp exposure. (l.bjorndal et al.2019).4.Vital tooth with signs and symptoms of mild and moderate pulpitis .Mild pulpitis Heightened and lengthened reaction to cold, warmth and sweet stimuli that can last up to 20 s but then subsides, possibly percussion sensitive. According to the histological situation that fits these findings, it would be implied that there is limited local inflammation confined to the crown pulp (W. J. Wolters et al.).Moderate pulpitis Clear symptoms, strong, heightened and prolonged reaction to cold, which can last for minutes, possibly percussion sensitive and spontaneous dull pain that can be more or less suppressed with pain medication. According to the histological situation that fits these findings, it would be implied that there is extensive local inflammation confined to the crown pulp.5.Occlusal pulp exposure because of caries removal.6.Exposure size upto 0.5 to 1 mm

-

Exclusion Criteria:

1.No pulp exposure after caries excavation.2.No bleeding after pulp exposure.3.The presence of a previous restoration of the tooth.4.Participants who not signed the written consent form.5.Patient with PAI score >2.

6.Severe pulpits-There are any clinical symptoms of Severe spontaneous pain and clear pain reaction to warmth and cold stimuli, often, sharp to dull throbbing pain, patients have trouble sleeping because of the pain (gets worse when lying down).7.Tooth is very sensitive to touch and percussion.

8.Evidence of internal or external resorption, calcified canals, as assessed by radiographic examination.9.Patients with periodontal disease, swelling and sinus tract.10.A positive history of antibiotic use within 1 month and analgesic use within week before the treatment.

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
1.Clinical success rate | [ baseline to 12 months]
  Clinical criteria of success:- 1.No pain or discomfort except for the first few days after treatment. 2.No tenderness to palpation or percussion and the tooth is functional. 3.Normal mobility and probing pocket depth. 4.Healthy soft tissues around teeth with no swelling, sinus tract.
2.Radiographic success rate | [Time Frame: baseline to 12 months]
  Radiographic success criteria:- 1.No pathosis such as root resorption, furcal pathosis or new periapical pathosis evident on the radiograph. 2.Complete radiographic healing

SECONDARY OUTCOMES:
3. Post Operative Pain | [Time Frame: Baseline to 7 days]]
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score100 means maximum pain. To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 100 millimeter line. Score 0 means no pain and Score 100 means maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: dr. sanjay tewari, Study Director — PGIDS, Rohtak, Haryana 124001
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code